CLINICAL TRIAL: NCT03282591
Title: A Randomized, Double-blind, Placebo-controlled Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Refractory Chronic Cough
Brief Title: Study of the Efficacy, Safety, and Tolerability of Serlopitant for the Treatment of Refractory Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTI-110; 2017-003250-16 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Results first posted 2019-10-22 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 5 mg Serlopitant Tablets (Experimental): Serlopitant Tablets
  Interventions: Drug: 5 mg Serlopitant Tablets
- Matching Placebo Tablets (Placebo Comparator): Placebo Tablets
  Interventions: Drug: Matching Placebo Tablets

INTERVENTIONS:
Drug: 5 mg Serlopitant Tablets — Serlopitant Tablets
  Other Names: VPD-737
  Arms: 5 mg Serlopitant Tablets
Drug: Matching Placebo Tablets — Placebo Tablets
  Arms: Matching Placebo Tablets

SUMMARY:
Study of the efficacy, safety, and tolerability of serlopitant for the treatment of refractory chronic cough

ELIGIBILITY:
Inclusion Criteria:

* Female and males between 18 and 80 years of age
* Have a diagnosis of treatment refractory chronic cough or unexplained cough for at least one year
* Chest radiograph or computed tomography (CT) Thorax within the last 5 years not demonstrating any abnormality considered to be significantly contributing to the chronic cough
* At Screening have a score of ≥ 40mm on the Cough Severity VAS
* At Baseline (Day 0) have a score of ≥ 40mm on the Cough Severity VAS
* All female subjects who are of childbearing potential must practice highly effective contraception (i.e., pregnancy prevention method with a failure rate of < 1% per year) from the time of the initial screening visit until 4 weeks after last dose of study drug. Please refer to the protocol for acceptable methods of contraception

Exclusion Criteria:

* Prior treatment with serlopitant or other NK1-R antagonist
* Presence of any medical condition or disability that could interfere with study
* History of hypersensitivity to serlopitant or any of its components
* Currently pregnant or male partner of pregnant female
* Females of childbearing potential who are unable or unwilling to use adequate contraception or who are breast feeding
* Current smoker or individuals who have given up smoking within the past 12 months
* FEV1/FVC < 60%
* Body mass index (BMI) <18 kg/m2 or ≥ 40 kg/m2 at Screening
* History of upper or lower respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Baseline Visit (Day 0)
* History of cystic fibrosis
* History of opioid use within 1 week of the Baseline Visit (Day 0)
* Requiring concomitant therapy with prohibited medications
* Treatment with biologic therapies within 8 weeks or 5 half-lives prior to the Baseline Visit (Day 0), whichever is longer
* Treatment with strong CYP3A4 inhibitors within 4 weeks prior to the Baseline Visit (Day 0)
* Treatment with any investigational therapy within 4 weeks (investigational biologic therapies within 8 weeks) prior to the Baseline Visit (Day 0)
* Serum creatinine, total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2x the upper limit of normal (ULN) during screening
* Positive test for any drug of abuse
* History of malignancy within 5 years prior to the Baseline Visit (Day 0), with the exception of completely treated and non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin
* Any known psychiatric diagnosis meeting DSM-5 criteria which may confound the assessment of serlopitant safety or efficacy, or interfere with the subject's ability to comply with protocol-mandated activities, within 3 years prior to randomization. Examples of such DSM-5 diagnoses include but are not limited to major depressive disorder, bipolar disorder, schizophrenia, psychotic disorder, intellectual disability, severe alcohol use disorder.
* Known active hepatitis infection
* Known history of human immunodeficiency virus (HIV) infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacky Smith, Principal Investigator — University of Manchester, United Kingdom
Locations (39):
- United States (29):
  - Study Site 130, Los Angeles, California
  - Study Site 128, Mission Viejo, California
  - Study Site 123, San Diego, California
  - Study Site 127, San Jose, California
  - Study Site 131, Stockton, California
  - Study Site 106, Colorado Springs, Colorado
  - Study Site 113, Colorado Springs, Colorado
  - Study Site 108, Denver, Colorado
  - Study Site 118, Largo, Florida
  - Study Site 107, Winter Park, Florida
  - Study Site 115, Plymouth, Minnesota
  - Study Site 110, Rochester, Minnesota
  - Study Site 121, Ocean Township, New Jersey
  - Study Site 125, Rochester, New York
  - Study Site 129, Charleston, North Carolina
  - Study Site 103, Charlotte, North Carolina
  - Study Site 111, Gastonia, North Carolina
  - Study Site 114, Mooresville, North Carolina
  - Study Site 122, Cincinnati, Ohio
  - Study Site 112, Tulsa, Oklahoma
  - Study Site 117, Eugene, Oregon
  - Study Site 116, Portland, Oregon
  - Study Site 104, Rock Hill, South Carolina
  - Study Site 102, Dallas, Texas
  - Study Site 120, Dallas, Texas
  - Study Site 101, San Antonio, Texas
  - Study Site 109, Waco, Texas
  - Study Site 126, Bellingham, Washington
  - Study Site 105, Greenfield, Wisconsin
- United Kingdom (10):
  - Study Site 133, Belfast
  - Study Site 139, Birmingham
  - Study Site 136, Cottingham
  - Study Site 141, Llanelli
  - Study Site 138, London
  - Study Site 137, London
  - Study Site 132, Manchester
  - Study Site 135, Oxford
  - Study Site 134, Preston
  - Study Site 140, Taunton

RESULTS

PARTICIPANT FLOW:
Groups:
- Serlopitant 5 mg: Subjects received a 3-tablet oral loading dose on the first day of the treatment period followed by a tablet taken once daily for 84 days.
- Placebo: Subjects received a 3-tablet Placebo loading dose on the first day of the treatment period followed by a tablet taken once daily for 84 days.
Period: Overall Study
Arm/Group | Serlopitant 5 mg | Placebo
Started | 92 | 93
Completed | 88 | 89
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: These figures represent the Full Analysis set (FAS) and is defined as all randomized subjects who received any amount of study treatment and had Baseline and at least one post baseline observation of the primary endpoint during the treatment period.
Groups:
- Placebo: Subjects received a 3-tablet oral loading dose on the first day of the treatment period followed by a tablet taken once daily for 84 days.
- Total: Total of all reporting groups
Arm/Group | Serlopitant 5 mg | Placebo | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.21) | 62.6 (10.09) | 62.6 (10.63)
Age, Continuous [Median (Full Range); unit: years] | 65.5 [28 to 79] | 64.5 [26 to 80] | 65 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 67 | 135
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 83 | 87 | 170
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 83 | 83 | 166
  More than one race | NA — This criterion was not collected. | NA — This criterion was not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 69 | 68 | 137
  United Kingdom | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Objective Cough Frequency (Log Normalized Percent Change Relative to Placebo)
Description: Change in 24-hour objective cough frequency is total number of cough events during the monitoring period (24-hour interval)/24 (Total duration (in hours) for the monitoring period) which is captured through sound recordings by a custom-built digital recording device (VitaloJAK, Vitalograph, Ltd).
Time Frame: from Baseline to Day 84
Measure: Least Squares Mean (Standard Error); unit: coughs/hr
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 88 | 88
coughs/hr | -0.18 (0.09) | -0.45 (0.08)
Statistical Analysis 1: Comparison: Serlopitant 5 mg vs Placebo; Test type: Superiority; p = 0.9942, Mixed Models Analysis; Mean Difference (Final Values) = 31.4, 95% CI 1-sided [upper limit 56.9]

2. Secondary Outcome: Change in Awake Objective Cough Frequency
Description: Awake cough frequency = (total number of cough events during the monitoring period (24-hour interval) the subject is awake)/(Total duration (in hours) for the monitoring period the subject is awake) which is captured by a custom-built digital recording device (VitaloJAK, Vitalograph, Ltd).
Time Frame: from Baseline to Day 84
Measure: Least Squares Mean (90% Confidence Interval); unit: coughs/hr
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 88 | 88
coughs/hr
  Day 28 (Week 4) | -0.12 [-0.26 to 0.01] | -0.30 [-0.43 to -0.17]
  Day 56 (Week 8) | -0.25 [-0.39 to -0.10] | -0.32 [-0.47 to -0.18]
  Day 84 (Week 12) | -0.19 [-0.34 to -0.04] | -0.46 [-0.60 to -0.31]

3. Secondary Outcome: Percentage of Participants With ≥ 30% Reduction in 24-hour Objective Cough Frequency
Description: The percentage of participants with ≥ 30% of reduction from baseline in 24-hour cough frequency is the number of participants with ≤-30% change in 24-hour cough frequency divided by the total number of participants with available data. This data is captured by a custom-built digital recording device (VitaloJAK, Vitalograph, Ltd).
Time Frame: from Baseline to Day 84
Measure: Number; unit: Percentage of participants
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 88 | 88
Percentage of participants | 71.4 | 90.2

4. Secondary Outcome: Percentage of Participants With ≥30% Reduction in Awake Objective Cough Frequency
Description: The percentage of participants with ≥ 30% of reduction from baseline in the awake cough frequency is the number of participants with ≤30% change in awake cough frequency divided by the total number of participants with available data. This data is captured by a custom-built digital recording device (VitaloJAK, Vitalograph, Ltd).
Time Frame: from Baseline to Day 84
Measure: Number; unit: percentage of participants
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 88 | 88
percentage of participants | 32.6 | 37.0

5. Secondary Outcome: Change From Baseline in Cough Severity Visual Analog Scale (VAS)
Description: Visual Analog Scale (VAS) 101-point scale ranging from 0 (no cough) to 100 (worst cough). A higher score corresponds to higher cough severity.
Time Frame: from Baseline to Day 84
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Serlopitant 5 mg | Placebo
Number analyzed (Participants) | 88 | 88
units on a scale
  Day 28 (Week 4) | -10.2 [-14.6 to -5.8] | -9.9 [-14.4 to -5.5]
  Day 56 (Week 8) | -14.6 [-19.4 to -9.8] | -7.4 [-12.3 to -2.5]
  Day 84 (Week 12) | -14.2 [-19.2 to -9.3] | -9.9 [-15.0 to -4.9]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were recorded from the first study drug administration through the follow-up visit at approximately Day 112 (± 3 days). After the Follow-Up visit, only SAEs that are believed to be drug related will be reported, without a specific end time.
Description: The at risk safety population is a subset of participants who received at least one dose of study medication. This population is analyzed based upon the actual treatment received, at the highest dose received.
Arm/Group | Serlopitant 5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 3/92 | 3/92
Other Adverse Events (participants affected / at risk) | 43/92 | 28/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=92) | Placebo (N=92)
Urosepsis (Infections and infestations) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serlopitant 5 mg (N=92) | Placebo (N=92)
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 6
Headache (Nervous system disorders) | 6 | 8
Urinary tract infection (Infections and infestations) | 6 | 3
Bronchitis (Infections and infestations) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Fatigue (General disorders) | 5 | 6
Dizziness (Nervous system disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Sinusitis (Infections and infestations) | 4 | 4
Acute sinusitis (Infections and infestations) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 2
Hypertension (Vascular disorders) | 3 | 0
Viral Upper respiratory tract infection (Infections and infestations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03282591/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03282591/SAP_001.pdf